CLINICAL TRIAL: NCT03195803
Title: Evaluation of Differential Effects of a Computer-based-cognitive Intervention on Cognition Among Elderly With Mild Cognitive Impairment With and Without White Matter Hyperintensities: A Comparative Study.
Brief Title: Cognitive Intervention in Mild Cognitive Impairment With or Without White Matter Hyperintensities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leila DJABELKHIR (Other)
Responsible Party: Sponsor-Investigator, Leila DJABELKHIR, PhD candidate, Broca Hospital
Organization: Broca Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LUS2WMH
Record Dates: First submitted 2017-06-14; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Comparison, non-randomized single blind study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCI with WMH (Experimental): Computerized Cognitive Stimulation was administered to this group, twice a week.
  Interventions: Behavioral: Computerized Cognitive Stimulation
- MCI without WMH (Active Comparator): Computerized Cognitive Stimulation was administered to this group, twice a week.
  Interventions: Behavioral: Computerized Cognitive Stimulation

INTERVENTIONS:
Behavioral: Computerized Cognitive Stimulation — All participants performed 12-week, 60-minutes twice a week of a computer-based cognitive stimulation program in group-setting, using a tablet with a software with specific training focused on attention, executive and speed processing functions.

SUMMARY:
This is a non-pharmacological study evaluating the differential effects of a computerized cognitive stimulation program according to the existence or not of white matter hyperintensities in elderly with mild cognitive impairment.

DETAILED DESCRIPTION:
White matter hyperintensities (WMH) are increasingly recognized as a factor determining the heterogeneity of Mild Cognitive Impairment (MCI) and have been associated to executive and processing speed impairment. Cognitive interventions in MCI remain quite limited for these MCI with vascular profile and studies often distinguish patients by clinical subtypes rather than brain profile before an intervention. Considering magnetic resonance imaging (MRI) data, this study investigated the effects of a computer-based cognitive stimulation (CCS) program on MCI with WMH compared to MCI without WMH.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Mild Cognitive Impairment
* With and without white matter hyperintensities
* MRI available or accept to perform one
* No engagement in other cognitive intervention program

Exclusion Criteria:

* Psychiatric and neurological disorders
* History of alcohol or other substance abuse
* Sensory and/or motor deficit affecting the use of a tablet

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Rey Auditory Verbal Learning test | Baseline assessment, change from Baseline on Rey Auditory Verbal Learning test at 3 months immediately after intervention and at 3 months follow-up
  Assessment of verbal learning in episodic memory

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie AR RIGAUD, Professor, Principal Investigator — Broca University Hospital

IPD SHARING:
Plan to Share IPD: No